CLINICAL TRIAL: NCT04672278
Title: A Randomized, Double-Blind, Placebo-Controlled Cross-Over Study to Evaluate the Safety, Lipid-Lowering Effect and Hypotensive Effect of Shanzha Fruit Drink in Patients With Mild to Moderate Hyperlipidemia
Brief Title: Lipid-Lowering Effect and Hypotensive Effect of Shanzha Fruit Drink in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Tomlinson, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BS/CR/PC/01
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hyperlipidemia; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Dietary Supplement: Shanzha Fruit drink or placebo drink
- Group B (Experimental)
  Interventions: Dietary Supplement: Shanzha Fruit drink or placebo drink

INTERVENTIONS:
Dietary Supplement: Shanzha Fruit drink or placebo drink — The dosage of Shanzha fruit drink or the placebo is 3 cans per day
  Other Names: placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, cross-over study. Subjects who meet the inclusion/exclusion criteria will be randomly and alternatively assigned to receive Shanzha fruit drink or placebo drink in the first 2 months or the last two months of the 5 months study period. In between the first and second treatment period, all patients will enter a Washout Period of 4 weeks and during which time patients should not receive any of the study functional fruit drink.

ELIGIBILITY:
Inclusion Criteria:

* • Total Cholesterol between 200-300 mg/dl (5.2-7.8 mmol/l).

  * Mean plasma triglyceride >= 4.5 mmol/l.
  * Diastolic blood pressure 95-100 mm Hg and/or Systolic blood pressure 130-150 mm Hg.
  * Be able to give written informed consent prior to study start and comply with study requirements.

Exclusion Criteria:

* • Total Cholesterol between 200-300 mg/dl (5.2-7.8 mmol/l).

  * Mean plasma triglyceride < 4.5 mmol/l.
  * Diastolic blood pressure 95-100 mm Hg and/or Systolic blood pressure 130-150 mm Hg.
  * Be able to give written informed consent prior to study start and comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the hypolipidemic effect of Shanzha Fruit drink in patients with hyperlipidemia | 5 months.
  The lipid profile including total cholesterol, HDL cholesterol, LDL-cholesterol and triglycerides will be measured at the start and the end of the study and changes from the baseline to the end of the treatment will be evaluated.
To evaluate the safety of Shanzha Fruit drink in patients with hyperlipidemia by monitoring of liver function tests. | 5 months.
  Alanine transaminase (ALT) levels as the main liver function test will be measured at the start and the end of the study.

SECONDARY OUTCOMES:
To evaluate the hypotensive effect of Shanzha Fruit Drink | 5 months.
  The changes in the systolic and diastolic blood pressure from the baseline to the end of the treatment will be evaluated.
To evaluate the safety of Shanzha Fruit drink in patients with hyperlipidemia by recording any adverse events reported by the study subjects or noted by the investigator. | 5 months.
  Any adverse events reported by the study subjects or noted by the investigator will be recorded at all the study visits after the initial study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No